CLINICAL TRIAL: NCT02779361
Title: Effect of Tea Consumption on Steroid Profile in Healthy Volunteers. Pilot Study
Brief Title: Effect of Tea Consumption on Steroid Profile in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: World Anti-Doping Agency (Other)
Responsible Party: Principal Investigator, Clara Pérez, PhD, Parc de Salut Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMIMFTCL/EGCG/3
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers; Doping in Sports
Keywords: green tea; steroid profile
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Green tea (Experimental): Green tea consumption along 7 days.
  Interventions: Dietary Supplement: Green tea

INTERVENTIONS:
Dietary Supplement: Green tea — Lipton pure green tea, 5 teas on the first 6 days, and 9 teas on the day 7. Teas will be ingested at 08:00 am, 10:30 am, 13:00 pm, 15:30 pm, 18:00 pm days 1-6, and 08:00 am (*), 10:30 am, 13:00 pm (*), 15:30 pm, 18:00 pm (*), 20:30 pm on day 7.
  One bag of tea will be used to prepare the beverages with exception of some beverages on day 7 that will be prepared with two bags (*).

SUMMARY:
Open label phase I clinical trial in healthy volunteers designed to assess changes on steroid profile after green tea consumption.

DETAILED DESCRIPTION:
Anabolic androgenic steroids are included in the list of banned substances in sports by the World Anti-Doping Agency (WADA) because of its ability to improve the performance of athletes.

Testosterone glucuronization by UGT2B17 isoenzyme (Uridine Diphosphate Glucuronyltransferase 2B17) is inhibited in vitro by green tea flavonols like epicatechin, epigallocatechin gallate (EGCG) and catechin gallate.

Therefore a diet rich in green tea could interfere in androgens' glucuronization and cause a change on the steroid profile of the athletes that could be considered a false positive.

A clinical trial designed to assess changes on steroid profile in healthy volunteers after green tea consumption will be conducted. Subjects with different UGT2B17 genotype will be recruited (10 of each type: ins/ins, ins/del, del/del) to study if the genotype can modulate the results obtained.

Urine samples obtained before and during 7 days of green tea consumption will be used to compare steroid profile. Blood samples will be also collected to assess EGCG pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Understand and accept the study's procedures and sign an informed consent form
* Body mass index (BMI=weight/heigth2) between 19 and 27 kg/m2, weight between 50 and 100 kg.
* No evidence of somatic or psychiatric disorders as per past medical history and physical examination
* EKG, blood and urine tests taken before entry into the study within the normal range. Minor and transient abnormalities may be acceptable if, according to the Principal Investigator's criterion and the state of the art, they are felt to have no clinical relevance, entail no danger to the participant, and don't interfere with the product's assessment. These abnormalities and their non-relevance must be specifically justified in writing)

Exclusion Criteria:

* Evidence of a preexisting condition (including gastrointestinal, liver, or kidney disorders) that may alter the absorption, distribution, metabolism or excretion of the drug or symptoms suggestive of drug-induced gastrointestinal irritation
* Previous psychiatric disorders, alcoholism, abuse of prescription drugs or illegal substances or regular consumption of psychoactive drugs
* Having donated blood or having participated in this same study in the preceding 8 weeks, or having participated in any clinical trial with drugs in the preceding 12 weeks
* Having had any somatic disease or having undergone major surgery in the 3 months prior to inclusion in the trial
* Individuals intolerant or having experienced a severe adverse reaction to green tea or caffeine
* Having regularly taken medication in the month before the trial, except for vitamins, herb-based remedies, dietary supplements that if, according to the Principal Investigator or his appointed collaborators' opinion, they pose no threat to the subjects and they won't interfere with the study's objectives. Single doses of symptomatic drugs taken during the week before the experimental session will not constitute an exclusion criterion if it can be assumed that it has been completely eliminated on the day of the experimental session
* Smokers of >10 cigarettes/day
* Consumption of >40 g/day of alcohol
* Daily consumption of less than one xanthine-containing beverages per day
* Hepatitis B, hepatitis C or human immunodeficiency virus-positive individuals
* Vegetarian subjects or with aberrant diets

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Steroid profile in urine | From 3 days before consumption (day -3,-2,-1) till day 8 (day 1-8) after consumption
  24 hours urine will be collected.

SECONDARY OUTCOMES:
Epigallocatechin gallate (EGCG) blood concentrations | Baseline and day 7
  One sample before tea administration (day -1) and 3 samples on day 7 (before, 1hour and 2 hours after first tea on day 7).
Serious and non serious adverse events | From inclusion till day 9 (final visit)
  Adverse events reported by subjects and interrogated by investigators will be collected.
UGT2B17 Genotype | Baseline
  Sample for pharmacogenetics will be obtained before tea administration

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Ventura, PhD, Study Director — World Anti-Doping Agency
Locations (1):
- Parc de Salut Mar-IMIM, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No